CLINICAL TRIAL: NCT02796833
Title: A Randomized Controlled Trial Comparing Two Commercially Available Lipid Emulsions in Patients Receiving Home Parenteral Nutrition - SMOF Versus Intralipid
Brief Title: Comparison of Two Intravenous Lipid Emulsions in Home Parenteral Nutrition Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johane Allard (Other)
Responsible Party: Sponsor-Investigator, Johane Allard, Professor of Medicine, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 14-8537-A
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Home Parenteral Nutrition
Keywords: Home parenteral nutrition; Liver injury; Intravenous Lipid Emulsions; Catheter-related infections; Safety
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMOF/Intralipid (Other): Patients that are randomized to receive for the first 6 months SMOF as a lipid emulsion in their PN, and for the next 6 month (after 28 days of active washout on Intralipid) Intralipid, which is the standard lipid emulsion used in the hospital. SMOF is approved by Health Canada.
  The parenteral nutrition bags are compounded individually for each patient based on their specific needs.
  Interventions: Drug: SMOFlipid20%
- Intralipid/SMOF (Other): Patients that are randomized to receive Intralipid, which is the standard lipid emulsion used in the hospital for the first 6 months, and for the next 6 month (after 28 days of active washout on Intralipid) SMOF as a lipid emulsion in their PN. SMOF is approved by Health Canada.The parenteral nutrition bags are compounded individually for each patient based on their specific needs.
  Interventions: Drug: SMOFlipid20%

INTERVENTIONS:
Drug: SMOFlipid20%

SUMMARY:
Total Parenteral Nutrition (TPN) is a way of feeding a person intravenously, and is required when the gastrointestinal tract is not able to function properly. TPN contains carbohydrates, protein, and fat and lipids. It also contains minerals and vitamins. The lipid that is currently used at the University Health Network home TPN program is Intralipid20%, which is based on Soybean oil, contains polyunsaturated fats and is a good source of energy and essential fatty acids, including omega 3 and 6 fatty acids, which needed by the body. However, long term use on Intralipid20% has been shown to have negative effects on antioxidant status, inflammation, liver, and the immune system.

SMOFlipid20% is a lipid emulsion that has been designed to maximize the ratio of omega 3 to omega 6 fatty acids, in an effort to avoid potentially harmful effects associated with Intralipid20%. In previous studies, it has been shown that SMOFlipid20% is safe and has positive benefits on the liver enzymes. There are no studies so far which follow patient who is on SMOFlipid20% long term. The investigators hope to show that with long term use of SMOFlipid20% is better for liver function compared to Intralipid20%.

DETAILED DESCRIPTION:
A prospective double-blind, crossover, randomized clinical trial of 13 months duration per participant to compare between 2 commercially available lipid emulsion, Intralipid vs SMOF, in patient receiving home parenteral nutrition (HPN). All subjects are stable HPN patients who receive Intralipid as lipid emulsion in their solutions. The subjects will be randomized to two groups. One group will receive Intralipid for 6 months, followed by 28 days of wash-out period, and then will receive SMOF for 6 months. Another groups will receive SMOF in first 6 months, followed by 28 days of wash-out period, then will receive Intralipid for 6 months. During wash-out period for both groups, the patients will receive Intralipid as standard lipid emulsion. Each patient will have 4 clinic visits at Toronto General Hospital for clinical interview, nutritional measurements, routine blood tests, and special blood tests at baseline then at 6, 7, 13 months. Also, the patients will be asked to have routine blood tests after month 3 and month 9. The patients will fill the food record which will be collected later after completion of each period, month 6 and 13 of the study. The investigators will be calling patients during both periods to check compliance and update on their condition including the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (ICF) to participate before any study related procedures are performed
* Adult over the age of 18
* Both males and females
* Clinically stable for at least 4 weeks with no acute medical co-morbidities
* Patients on a stable Intralipid HPN regimen for 6 months and expected to require long-term PN for at least 13 more months

Exclusion Criteria:

Subjects not already on Intralipid PN Inability to give informed consent Alcohol or drug abuse Pregnant and lactating women

Clinical instability such as the following:

* Acute pulmonary edema
* Decompensated heart failure
* Decompensated chronic liver disease
* Severe post-traumatic conditions
* Uncontrolled diabetes mellitus
* Acute myocardial infarction
* Acute stroke
* Acute thromboembolism
* Metabolic acidosis
* Sepsis
* Hypotonic dehydration
* Coagulopathy with prolonged aPTT or INR Elevated triglyceride level: more than 4.5 mmol/L Active malignancy with life expectancy less than one year Subjects who are hypersensitive or allergic to the product ingredients of SMOF or Intralipid, including soybean oil, peanuts, fish oil, and egg as well as allergy to peanuts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
change in alanine transaminase (ALT) | baseline 1, 6 months, baseline 2 (7 mo), 13 months

SECONDARY OUTCOMES:
changes in liver function tests (total and conjugated bilirubin, ALP, AST, GGT) | baseline 1, 6 months, baseline 2 (7 mo), 13 months
rate of infections (central line and other) per 1000 catheter days | baseline 1, 6 months, baseline 2 (7 mo), 13 months
antibiotic days for acute infections | baseline 1, 6 months, baseline 2 (7 mo), 13 months
number of hospitalizations for the past 6 months | baseline 1, 6 months, 13 months
number of catheter changes for the past 6 months | baseline 1, 6 months, 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Johane Allard, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clermont-Dejean NM, Schwenger KJP, Arca C, Somlaw N, Alhanaee A, Hortencio TDR, Jin J, Jung H, Lou W, Ma D, Allard JP. Comparing mixed oil to soybean oil lipid emulsion in patients on home parenteral nutrition: a pilot prospective double-blind, crossover, randomized trial. Pilot Feasibility Stud. 2023 Apr 20;9(1):64. doi: 10.1186/s40814-023-01295-1. PMID 37081524